CLINICAL TRIAL: NCT00970775
Title: A Phase I, Single Centre, Double-blind, Randomised, Placebo-controlled, Parallel-group Study to Assess the Safety, Tolerability and Pharmacokinetics of Oral AZD2423 After Single Ascending Doses in Healthy Japanese Male and Non-Fertile Female Volunteers
Brief Title: AZD2423 Single Ascending Dose Study in Healthy Japanese Subjects
Acronym: JSAD
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: MSD, AstraZeneca
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: D2600C00003
Record Dates: First submitted 2009-09-01; First posted 2009-09-02 (Estimated); Last update posted 2010-03-18 (Estimated); Status verified 2010-03

CONDITIONS: Healthy Volunteer
Keywords: Phase I; Japanese healthy volunteer; AZD2423

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1. AZD2423 (Experimental)
  Interventions: Drug: AZD2423
- 2. Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AZD2423 — oral solution, single dose
  Arms: 1. AZD2423
Drug: Placebo — oral solution,single dose
  Arms: 2. Placebo

SUMMARY:
This is a Phase I, single centre, randomised, double-blind, placebo-controlled, parallel group study to assess the safety, tolerability and pharmacokinetics of AZD2423 following single ascending dose administration to healthy Japanese subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Japanese male and non-fertile female subjects aged ≥20 to ≤55 years with suitable veins for cannulation or repeated venepuncture.
* Body weight 45-90 kg and Body mass index (BMI) ≥18.0 and ≤27.0 kg/m2
* Clinically normal physical findings including supine blood pressure, pulse rate, orthostatic blood pressure, ECG, and laboratory assessments in relation to age, as judged by the Investigator.

Exclusion Criteria:

* History of any clinically significant disease or disorder which, in the opinion of the Investigator, may either put the subject at risk because of participation in the study, or influence the results or the subject's ability to participate in the study.
* Any clinically significant illness/infection or medical/surgical procedure or trauma, as judged by the Principal Investigator, within 3 months of the first administration of investigational product.
* Frequent use of tobacco or other nicotine containing products. Frequent use is defined as smoking or consumption/intake of nicotine products more than two days per week during the last 12 weeks.

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2009-08; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
To asses the safety: Adverse events, vital signs, electrocardiograms (ECGs), laboratory variables. | From screening period to follow-up visit, 40 days (Maximum).

SECONDARY OUTCOMES:
To characterize the pharmacokinetics of AZD2423 in plasma and urine. | Blood and urine sampling from pre-dose until follow-up visit, 10 days (approximately)
Exploratory endpoints;Levels of CCL2 pre-and post dose | Blood sampling after dosing, 3 days

CONTACTS AND LOCATIONS:
Overall Officials: Ulrike Lorch, MD MFPM FRCA, Principal Investigator — Richmond Pharmacology Limited
Locations (2):
- United Kingdom (2):
  - Research Site, Croydon
  - Research Site, London